CLINICAL TRIAL: NCT02008682
Title: The Efficacy and Safety of Liraglutide Compared to Sitagliptin, Both in Combination With Metformin in Chinese Subjects With Type 2 Diabetes.(LIRA-DPP-4 CHINA™)
Brief Title: The Efficacy and Safety of Liraglutide Compared to Sitagliptin, Both in Combination With Metformin in Chinese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN2211-4075; U1111-1139-0016 (Other: WHO)
Record Dates: First submitted 2013-12-05; First posted 2013-12-11 (Estimated); Results first posted 2015-12-22 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide 1.8 mg + metformin (Experimental): 2-week screening period, 26-week treatment duration, and a 1-week follow-up period
  Interventions: Drug: liraglutide
- Sitagliptin 100 mg + metformin (Active Comparator): 2-week screening period, 26-week treatment duration, and a 1-week follow-up period
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: liraglutide — Administered subcutaneously (s.c., under the skin) once daily as add-on to the subject's stable pre-trial metformin dose.
  Arms: Liraglutide 1.8 mg + metformin
Drug: sitagliptin — Administered orally once daily as add-on to the subject's stable pre-trial metformin dose.
  Arms: Sitagliptin 100 mg + metformin

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to investigate the efficacy and safety of liraglutide compared to sitagliptin, both as add-on to metformin in Chinese subjects with type 2 diabetes inadequately controlled on metformin monotherapy. Eligible subjects will continue their metformin background treatment during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age at least 18 years and below 80 years at the time of signing informed consent
* Subjects diagnosed type 2 diabetes mellitus and treated with metformin monotherapy at a stable dose of at least 1500 mg daily or maximum tolerated dose above or equal to 1000 mg daily for at least 60 days prior to screening
* HbA1c 7.0-10.0% (both inclusive)
* Body mass index below or equal to 45.0 kg/m^2

Exclusion Criteria:

* Treatment with glucose lowering agent(s) other than stated in the inclusion criteria in a period of 60 days prior to screening. An exception is short-term treatment (below or equal to 7 days in total) with insulin in connection with intercurrent illness
* History of chronic pancreatitis or idiopathic acute pancreatitis
* Any chronic disorder or severe disease which at the discretion of the investigator might jeopardise subject's safety or compliance with the protocol
* Screening calcitonin value above or equal to 50 ng/l
* Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2
* Diagnosis of malignant neoplasm in the previous 5 years (except basal cell skin cancer or squamous cell skin cancer)
* Any contraindications to liraglutide, sitagliptin or metformin according to local labelling

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (16):
- China (16):
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Cangzhou, Hebei
  - Novo Nordisk Investigational Site, Hengshui, Hebei
  - Novo Nordisk Investigational Site, Shijiazhuang, Hebei
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Suzhou, Jiangsu
  - Novo Nordisk Investigational Site, Wuxi, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Dalian, Liaoning
  - Novo Nordisk Investigational Site, Shenyang, Liaoning
  - Novo Nordisk Investigational Site, Qingdao, Shandong
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Beijing

REFERENCES:
- [Result] Zang L, Liu Y, Geng J, Luo Y, Bian F, Lv X, Yang J, Liu J, Peng Y, Li Y, Sun Y, Bosch-Traberg H, Mu Y. Efficacy and safety of liraglutide versus sitagliptin, both in combination with metformin, in Chinese patients with type 2 diabetes: a 26-week, open-label, randomized, active comparator clinical trial. Diabetes Obes Metab. 2016 Aug;18(8):803-11. doi: 10.1111/dom.12674. Epub 2016 May 20. PMID 27060930
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 25 sites in China.
Pre-assignment Details: Between screening and randomisation, eligible subjects were to continue their usual pre-trial metformin dose and dosing frequency.
Groups:
- Liraglutide: subcutaneously, once-daily dose of liraglutide 1.8 mg with metformin at pre-trial stable dose (at least 1500 mg or maximum tolerated dose at least 1000 mg daily). Liraglutide dose was escalated from 0.6 mg/day to 1.8 mg/day during 3-4 weeks.
- Sitagliptin: orally, once-daily dose of sitagliptin 100 mg with metformin at pre-trial stable dose (at least 1500 mg or maximum tolerated dose at least 1000 mg daily).
Period: Overall Study
Arm/Group | Liraglutide | Sitagliptin
Started | 184 | 184
Exposed | 183 (1 subject withdrawn before exposure to trial product) | 184
Completed | 157 (Completed without discontinuation of trial product) | 170 (Completed without discontinuation of trial product)
Not Completed | 27 | 14

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all subjects receiving at least one dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide | Sitagliptin | Total
Number analyzed (Participants) | 183 | 184 | 367
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.7) | 51.4 (11.0) | 51.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 67 | 148
  Male | 102 | 117 | 219
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.32 (3.389) | 27.16 (4.029) | 27.24 (3.720)
Body weight [Mean (Standard Deviation); unit: kg] | 76.17 (13.562) | 75.78 (15.089) | 75.98 (14.330)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 5.31 (4.39) | 5.22 (5.40) | 5.27 (4.92)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.26 (2.216) | 9.46 (2.237) | 9.36 (2.226)
Glycosylated haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin] | 8.14 (0.833) | 8.11 (0.780) | 8.12 (0.806)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Haemoglobin (HbA1c)
Description: Mean change from baseline in glycosylated haemoglobin A1c (HbA1c) at Week 26.
Time Frame: Week 0, week 26
Population: Full analysis set was defined as all randomised and exposed subjects who had any post randomisation data. Missing data was imputed using a mixed model for repeated measurements. The subjects would not contribute to the analyses if they didn't have a corresponding post-baseline value.
Measure: Mean (Standard Deviation); unit: Percent (%) glycosylated haemoglobin
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 162 | 175
Percent (%) glycosylated haemoglobin | -1.666 (0.9982) | -0.969 (0.9742)

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Mean change from baseline in fasting plasma glucose (FPG) at Week 26.
Time Frame: Week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 168 | 180
mmol/L | -2.347 (2.1655) | -1.205 (2.2961)

3. Secondary Outcome: Change From Baseline in 7-point Self-measured Plasma Glucose Profile
Description: Mean change from baseline in mean of 7-point self-measured plasma glucose at week 26. The 7-point self-measured plasma glucose levels were measured before and after (120 minutes after the start of the meal) the three main meals (breakfast, lunch and dinner), and at bed time.
Time Frame: Week 0, week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 161 | 174
mmol/L | -2.25 (2.244) | -1.36 (2.204)

4. Secondary Outcome: Subjects Who Achieve (Yes/no) HbA1c Below 7.0 % (American Diabetes Association Target)
Description: Calculated as the percentage of subjects achieving treatment target of HbA1c < 7.0% at Week 26
Time Frame: After 26 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 162 | 175
percentage of subjects | 76.5 | 52.6

5. Secondary Outcome: Subjects Who Achieve (Yes/no) HbA1c Below or Equal to 6.5 % (American Association of Clinical Endocrinologists Target)
Description: Calculated as the percentage of subjects achieving treatment target of HbA1c <= 6.5% at Week 26
Time Frame: After 26 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 162 | 175
percentage of subjects | 61.7 | 26.3

6. Secondary Outcome: Number of Confirmed Hypoglycaemic Episodes
Description: confirmed hypoglycaemic episode defined as severe (unable to treat her/himself) or biochemically confirmed by a plasma glucose < 3.1 mmol/L
Time Frame: Weeks 0-26
Population: Safety analysis set included all subjects receiving at least one dose of investigational product.
Measure: Number; unit: episodes
Arm/Group | Liraglutide | Sitagliptin
Number analyzed (Participants) | 183 | 184
episodes | 2 | 1

ADVERSE EVENTS:
Time Frame: Weeks 0-26
Description: Treatment emergent adverse event defined as an event that had onset date (or increase in severity) on or after the first day of exposure to trial product and no later than seven days after the last day of trial product. Safety analysis set defined as all exposed subjects.
Arm/Group | Liraglutide | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 3/183 | 6/184
Other Adverse Events (participants affected / at risk) | 65/183 | 14/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=183) | Sitagliptin (N=184)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thymoma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (N=183) | Sitagliptin (N=184)
Nausea (Gastrointestinal disorders) | 27 (30) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 15 (16) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 20 (20) | 1 (1)
Lipase increased (Investigations) | 11 (11) | 8 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.